CLINICAL TRIAL: NCT06656520
Title: Impact of Telehealth Care on Clinical Outcomes in Heart Failure Patients
Brief Title: Impact of Telehealth Care
Status: Withdrawn | Type: Observational
Why Stopped: A retrospective observational study was conducted using electronic medical record data
Sponsor: Pei-Hung Liao (Other)
Collaborators: Mackay Memorial Hospital (Other); National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Pei-Hung Liao, Professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Other Study IDs: 23MMHIS219e
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Telehealth Services; Telehealth
Keywords: Telehealth, heart failure, rehospitalization, mortality
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure is associated with high incidence and mortality rates, limited physical activity, decreased quality of life, and increased healthcare expenses. Implementing a Telehealth Care (TC) HF program could address these challenges while improving patient outcomes.

DETAILED DESCRIPTION:
Telemonitoring for heart failure patients reduces all-cause and cardiovascular mortality by enabling early intervention during clinical deterioration, improving outcomes even for those recently discharged. Moreover, a reduction in the percentage of days lost due to unplanned cardiovascular hospital admissions is evident. Furthermore, the rapid expansion of telehealth care and telemedicine services during the COVID-19 pandemic optimized the management and care quality of heart failure patients through telemonitoring .

ELIGIBILITY:
Inclusion Criteria:

* Inpatients diagnosed with heart failure were enrolled, with patients automatically selected daily by the electronic medical record system. A list of ward visits was obtained based on the first three digits of the International Classification of Diseases 10th edition diagnosis codes; the ICD-10 code I50 was applied for selection.

Exclusion Criteria:

* Other diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients diagnosed with heart failure were enrolled, with patients automatically selected daily by the electronic medical record system. A list of ward visits was obtained based on the first three digits of the International Classification of Diseases 10th edition diagnosis codes; the ICD-10 code I50 was applied for selection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
mortality and rehospitalization rates | After discharge one year
  analyze the one-year all-cause mortality and rehospitalization rates in patients with and without telehealth care while examining cardiovascular mortality and rehospitalization rates simultaneously.

IPD SHARING:
Plan to Share IPD: No